CLINICAL TRIAL: NCT02177682
Title: An Open-label, Dose Escalation, Phase I Study to Evaluate the Tolerability, Safety and Pharmacokinetics of Afuresertib Monotherapy in Japanese Relapsed Multiple Myeloma Patients.
Brief Title: Study of Afuresertib Monotherapy in Japanese Relapsed Multiple Myeloma Patients
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115960
Record Dates: First submitted 2014-05-29; First posted 2014-06-30 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Neoplasms, Haematologic
Keywords: AKT inhibitor; Afuresertib; multiple myeloma
MeSH Terms: conditions — Neoplasms; Multiple Myeloma | interventions — afuresertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Afuresertib (Experimental): Three subjects will be enrolled and given afuresertib 125 mg orally and monitored for toxicity. After completion of PK sampling in 3 days (Cycle 0), daily repeated dose of 125 mg will be given for 21 days (Cycle 1). If no DLT event is found after 21 days of repeated dosing, up to 6 subjects will be enrolled and given afuresertib 150 mg. If afuresertib 150 mg is assessed to be tolerable, up to 6 subjects can be enrolled and given afuresertib 200 mg. If afuresertib 200 mg is assessed to be intolerable, up to 6 subjects will be enrolled and given afuresertib 150mg or 175 mg. In any Dose levels, if DLT occurs in more than 2 subjects, that Dose level will be considered as intolerable."
  Interventions: Drug: Afuresertib

INTERVENTIONS:
Drug: Afuresertib — Size 4 and Size 1 opaque white capsules containing 25 mg and 100 mg of afuresertib, respectively, to be administered orally.

SUMMARY:
Afuresertib, an AKT inhibitor, has shown in vitro and in vivo activity in multiple myeloma models. AKT inhibitor has also demonstrated encouraging clinical activity in multiple myeloma. This study is designed to determine the tolerability, safety, pharmacokinetics and efficacy of afuresertib as monotherapy in Japanese relapsed multiple myeloma patients. This is an open label, dose-escalating, phase I study. Afuresertib will be given daily until the subjects meet any study treatment withdrawal criteria including disease progression. A total of up to 24 subjects will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is provided.
* Japanese females or males aged 20 years or older (at the time consent is obtained).
* Histologically confirmed diagnosis of relapsed multiple myeloma.
* Performance score of 0 and 1 according to the ECOG scale.
* Relapsed after at least 1 line of systemic therapy. The preparative regimen (with or without total body irradiation) and subsequent autologous stem cell rescue used for an autologous stem cell transplant are considered as one line of therapy.
* Able to swallow and retain oral medication.
* Male subjects with a female partner of childbearing potential must have had a prior vasectomy or agree to use adequate contraception from the time of the first dose of study drug until three months after the last dose of study drug.
* A female subject is eligible to participate if she is of: (A) Non-childbearing potential (i.e. physiologically incapable of becoming pregnant): Pre-menopausal females with a documented tubal ligation or hysterectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea [if unclear, simultaneous follicle stimulating hormone >40 milli-international units (MIU)/milliliter (mL) and oestradiol <40 picograms (pg)/mL (<140 picomoles [pmol]/L) is required as confirmation]. (B) Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt must discontinue HRT to confirm post-menopausal status prior to study enrolment. Following confirmation, they can resume HRT during the study without use of a contraceptive method. (C) Child-bearing potential, has a negative serum pregnancy test within 7 days prior to enrolment, and agrees to use adequate contraception from screening until four weeks after the last dose of study drug. Note: The recommended contraceptive methods are abstinence of sexual intercourse, use of intrauterine device/system, vasectomy, and use of condom with spermicidal agent. An oral contraceptive drug does not offer a reliable contraceptive method as a drug-drug interaction may occur.
* Adequate organ system functions as defined in the protocol
* Subjects with a history of autologous stem cell transplant are eligible provided the following criteria are met: transplant completed >180 days prior to enrolment; no active infection (e.g. cytomegalovirus, varicella-zoster virus); meets the remainder of the eligibility criteria outlined in this protocol.

Exclusion Criteria:

* Chemotherapy, radiotherapy, immunotherapy or other anti-myeloma therapy within 28 days prior to enrolment. In addition, any toxicity (except alopecia) should be recovered to <=Grade 1 by National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 4.0.
* Use of an investigational drug within 30 days or five half-lives, whichever is longer.
* History of an allogenic stem cell transplant. For patients with history of autologous stem cell transplant, inclusion criteria 10 must be met.
* History of PI3K/AKT inhibitors.
* Current use of prohibited medication or subject who requires any of these medications during treatment of afuresertib, as well as subject who cannot meet the protocol specified meals and dietary restrictions
* Current use of oral corticosteroids, except inhaled or topical use.
* Uncontrolled diabetes mellitus by diet, exercise or medicinal therapies including insulin, and with fasting serum glucose >=130 mg/dL (>=7.28 millimoles [mmol]/L).
* Use of anticoagulants other than low dose (prophylactic) anticoagulants for subject whose Prothrombin time (PT)/international normalization ratio (INR) and activated partial thromboplastin time (APTT) is <=1.5 x upper limit of normal (ULN).
* Presence of active Gastro-intestinal (GI) disease or other condition that could affect GI absorption (e.g. malabsorption syndrome) or predispose subject to GI ulceration.
* Any major surgery that required hospitalization within last four weeks.
* Any serious or unstable pre-existing medical, psychiatric, or other conditions (including lab abnormalities) that could interfere with subject safety or obtaining informed consent.
* Active infection requiring parenteral or oral anti-infective treatment.
* Evidence of severe or uncontrolled systemic diseases (e.g., unstable or uncompensated respiratory, hepatic, renal, or cardiac disease).
* Central nervous system malignancies, primary or metastatic.
* Diagnosis of or treatment history for another malignancy within 2 years, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* History of known infection with human immunodeficiency virus (HIV).
* Positive hepatitis B surface (HBs) antigen or hepatitis B virus (HBV) Deoxyribonucleic acid (DNA). If negative for HBs antigen and positive for both or either of hepatitis B core (HBc) and HBs antibodies, HBV DNA needs to be negative.
* Positive hepatitis C virus (HCV) antibody
* Corrected QT interval (QTc) >450 milliseconds (msec) or QTc > 480 msec for patients with bundle branch block. The QTc is the QT interval corrected for heart rate according to Fridericia's formula (QTcF). Note: The QTc should be based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period.
* Other clinically significant ECG abnormalities, including 2nd or 3rd degree atrioventricular block.
* History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty or stenting or bypass grafting within the past six months.
* Class III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Pregnant or lactating female.
* Known hypersensitivity to any components of the study treatment.
* Others who are considered as inappropriate to participate in this study by investigators.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-08-13 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Dose-limiting toxicities (DLTs) when afuresertib is given as monotherapy | Day 1 to 21 of Cycle 1
  DLT is defined as an adverse event which is applicable to any of the criteria specified in the protocol and judged to have a reasonable causal relationship with afuresertib. The DLT evaluation period will be from the day of the first dosing in Cycle 1 to Day 21 of Cycle 1 or the day of DLT occurrence if any DLT occurred before Day 21 of Cycle 1.

SECONDARY OUTCOMES:
Eastern Cooperative Oncology Group (ECOG) performance status (PS) | From Day -3 until 30 days after the last dose of afuresertib
  The performance status will be assessed using the ECOG scale
Vital signs assessment | From Day -3 until 30 days after the last dose of afuresertib
  Vital sign measurements will include systolic and diastolic blood pressure and pulse rate
Number of participants with adverse events (AEs) | From Day -3 until 30 days after the last dose of afuresertib
  An AE is defined as any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Laboratory assessments | From Day -3 until 30 days after the last dose of afuresertib
  laboratory assessments will include haematologic tests, blood chemistry tests, coagulation tests, urine tests and lipid panel
12-lead electrocardiogram (ECG) assessment | From Day -3 until 30 days after the last dose of afuresertib
  Triple 12-lead ECGs will be obtained at designated time points during the study using an ECG machine that automatically calculates the heart rate and measures pulse rate (PR), QRS, QT, and QTc intervals.
Left ventricular ejection fraction (LVEF) assessment | From Day -3 until 30 days after the last dose of afuresertib
  Echocardiogram and/or Multi-gated Acquisition (MUGA) scans will be performed for evaluation for LVEF
Composite of pharmacokinetic (PK) parameters of afuresertib monotherapy administered as single and repeated dose | Cycle 0 (Pre-dose, 0.5 hour [hr],1 hr, 2 hr, 3 hr, 4hr, 6 hr, 8 hr, 24 hr, 48 hr, 72 hr) and Cycle 1 Day 8 (Pre-dose, 0.5 hr,1 hr, 2 hr, 3 hr, 4hr, 6 hr, 8 hr, 24 hr)
  PK parameters will include area under the concentration-time curve from time zero extrapolated to infinite time [AUC (0-infinity)], area under the concentration-time curve over the dosing interval [AUC (0-tau)], maximum observed plasma concentration (Cmax), last observed quantifiable concentration (Clast), apparent clearance following oral dosing (CL/F), pre-dose (trough) concentration at the end of the dosing interval (Ctau), time of occurrence of Cmax (tmax), terminal phase half-life (t1/2), steady state ratio (Rs) and observed accumulation ratio (Ro)
Response rate and clinical benefit rate (rate of minor response or better) | Within 4 weeks of Day 1 Cycle 1, at start of each cycle (except Cycle 1), and then every 6 to 9 weeks until 30 days after the last dose of afuresertib
  Response evaluations will be determined according to the Response Criteria for multiple myeloma as stringent complete response (sCR), complete response (CR), very good partial response (VGPR), partial response (PR), and minor response (MR). Response rate will be defined as the percentage of subjects with sCR, CR, VGPR or PR. Subjects with unknown or missing response will be treated as non-responder.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Japan (5):
  - Novartis Investigative Site, Aichi
  - Novartis Investigative Site, Fukuoka
  - Novartis Investigative Site, Miyagi
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Tokyo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17649